CLINICAL TRIAL: NCT03348111
Title: Establishing a New Protocol for Early Mucositis and Peri-implantitis Treatment Using an Air-polishing Device
Acronym: PERIFLOW
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No participant enrolled
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RC31/15/7854; 2016-A00754-47 (Other: ID-RCB)
Record Dates: First submitted 2017-10-30; First posted 2017-11-20 (Actual); Last update posted 2020-08-26 (Actual); Status verified 2020-08

CONDITIONS: Peri-Implantitis; Mucositis
Keywords: Mucositis; Peri-Implantitis; Air-Flow Master Piezon®
MeSH Terms: conditions — Peri-Implantitis; Mucositis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Air-polishing device (Experimental): Air polishing of the implant surface and/or elimination of the intrapocket biofilm using the air abrasion device Air-Flow Master Piezon®
  Interventions: Device: Air-polishing device

INTERVENTIONS:
Device: Air-polishing device — Air abrasion using the Air-Flow Master Piezon® with erythritol and Chlorhexidine powders on implants presenting clinical and radiographic signs of mucositis and peri-implantitis along with renewal of local oral hygiene instructions in order to reduce the inflammation locally
  Other Names: Air-Flow Master Piezon®

SUMMARY:
Considering the frequent occurence of peri-implantitis and mucositis, a multiple of treatment alternatives have been proposed including non-surgical and surgical procedures. However, it seems that the most effective treatment remains prevention of these diseases.

The aim of this study is to emphasize on mucositis and peri-implantitis prevention using an air abrasion device the Air-Flow Master Piezon® with erythritol and chlorhexidine powder in order to eliminate and / or disorganize the biofilm responsible for peri-implant mucosa inflammation.

DETAILED DESCRIPTION:
Peri-implant infections (mucositis and peri-implantitis) depict an increasing focus in dental practice and implantology. mean prevalence of mucositis is of 43% and periimplantitis of 22%. Consequences for the implant without successful treatment range from local reversible inflammation (mucositis) to implant loss (periimplantitis). These lead to functional, social and esthetic prejudices for patients. The main factor for establishment of peri-implant infections is the formation and maturation of the bacterial biofilm. Peri-implantitis and mucositis treatment require the removal of the bacterial biofilm and the disinfection of the implant surface. Because of special surface conditions and structures, it is more difficult to remove bacterial biofilms from implant surfaces than teeth. the key to controlling the inflammation due to the bacterial biofilm is to prevent its installation and progression. The procedure tested in this study is an air abrasion device, the Air-Flow Master Piezon® with erythritol and chlorhexidine powders on implants presenting clinical and radiographic signs of mucositis and peri-implantitis along with renewal of local oral hygiene instructions in order to reduce the inflammation locally by disorganizing and eliminating the biofilm. Follow-up of the patients will be held every 2 months for 6 months by scoring the bleeding on probing, the plaque index and measuring clinical attachment level in order to compare it with the initial measure. At 6 month an X-ray will also enable to compare bone level and mineralization. This initial study will help establish a standardized protocol for peri-implant infection management.

ELIGIBILITY:
Inclusion Criteria:

* adult patients,
* possessing one or more implants prosthetically engaged with local peri-implant mucosa inflammation assessed by bleeding on probing
* affiliated with a social security scheme

Exclusion Criteria:

* patients with implant mobility or implants associated with vestibular cellulitis
* not available patients for the follow-up visits
* patients with known allergy to erythritol and/or Chlorhexidine powder
* patients with chronic bronchitis
* patients with asthma
* patients with endocarditis
* patients with contagious disease
* patients with immunodeficiency
* patients under radiotherapy and/or chemotherapy and/or antibiotics
* not mastery of plaque control on the part of the patient (after education)
* subjects under legal protection
* pregnant or breastfeeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-06 (Estimated); Primary Completion 2021-06 (Estimated); Study Completion 2021-06 (Estimated)

PRIMARY OUTCOMES:
Change from baseline peri-implant inflammation at 6 months | 6 months
  bleeding on probing (binary criteria : yes/no)
Change from baseline peri-implant inflammation at 4 months | 4 months
  bleeding on probing (binary criteria : yes/no)
Change from baseline peri-implant inflammation at 2 months | 2 months
  bleeding on probing (binary criteria : yes/no)

SECONDARY OUTCOMES:
stability of the bone level | 6 months
  bone level assessed by X-ray
clinical attachment gain | 2 months
  The measurement of the probing depth and of the eventual recession (compared to Baseline) allows to assess the clinical attachment gain
clinical attachment gain | 4 months
  The measurement of the probing depth and of the eventual recession (compared to Baseline) allows to assess the clinical attachment gain
clinical attachment gain | 6 months
  The measurement of the probing depth and of the eventual recession (compared to Baseline) allows to assess the clinical attachment gain
Quality of life with Oral Health Assessment Tool (OHAT) | 6 months
  The Oral Health Assessment Tool (OHAT) was a component of the Best Practice Oral Health Model for Australian Residential Care study. The OHAT provided institutional carers with a simple, eight category screening tool to assess residents' oral health, including those with dementia
Quality of life with the Geriatric Oral Health Assessment Index (GOHAI) | 6 months
  The Geriatric Oral Health Assessment Index (GOHAI) is a self-reported measure designed to assess the oral health problems of older adults

CONTACTS AND LOCATIONS:
Overall Officials: Sara Laurencin, MD, Principal Investigator — University Hospital of Toulouse
Locations (1):
- University Hospital Toulouse (Faculty of Dental Surgery), Toulouse, France

IPD SHARING:
Plan to Share IPD: No